CLINICAL TRIAL: NCT07157202
Title: Association Between Helicobacter Pylori Infection and Disease Activity in Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: Associating Gastric Infection With Autoimmune Flare Severity in an Egyptians
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Wanees Ebrahim, resident at the Internal Medicine department, Assiut University
Other Study IDs: H. pylori and SLE
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: H. Pylori; SLE - Systemic Lupus Erythematosus
Keywords: SLE; H. pylori infection
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult patients with a confirmed diagnosis of SLE,: Eligible participants are adults (at least 18 years old) diagnosed with SLE according to ACR or SLICC criteria, who have not used antibiotics or proton pump inhibitors in the past four weeks, and provide written informed consent . Of those eligible, the expected sample size is 115 patients, calculated to power the main outcome analysis.

SUMMARY:
A cross-sectional, observational study aims to evaluate the relationship between Helicobacter pylori infection and disease activity in patients diagnosed with systemic lupus erythematosus (SLE), using a combination of structured patient interviews, standardized disease assessments, and laboratory detection of H. pylori by stool antigen testing .

DETAILED DESCRIPTION:
the study explores the potential role of chronic H. pylori infection as a trigger or aggravating factor in SLE, an autoimmune disorder characterized by overactive immune responses that cause multisystem organ damage . The rationale is based on recent findings suggesting that chronic infections may worsen autoimmune disease activity by persistent immune stimulation and production of cross-reactive autoantibodies . SLE patients attending clinics at Assiut University Hospital will be assessed over one year; inclusion requires confirmed SLE diagnosis per established criteria, absence of recent antibiotics/PPIs, and consent. Clinical data, disease activity (via SLEDAI-2K), and socio-demographic information will be collected through detailed medical interviews and laboratory investigations, particularly focusing on stool-based antigen tests for H. pylori. All data will be securely recorded for statistical analysis assessing the bidirectional impact of infection status and SLE severity .

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged ≥18 years) with a confirmed diagnosis of SLE according to the American College of Rheumatology (ACR) or Systemic Lupus International Collaborating Clinics (SLICC) classification criteria.

Patients who provide written informed consent to participate in the study. Patients who have not received antibiotics or proton pump inhibitors (PPIs) in the four weeks

Exclusion Criteria:

* Patients with a history of gastric surgery or known gastrointestinal malignancy.

  * Patients currently receiving immunosuppressive therapy for conditions other than SLE.
  * Patients with coexisting autoimmune diseases other than SLE.
  * Pregnant or lactating women.
  * Patients with active infections (other than H. pylori) at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants are adults (at least 18 years old) diagnosed with SLE according to ACR or SLICC criteria, who have not used antibiotics or proton pump inhibitors in the past four weeks, and provide written informed consent . Patients with prior gastric surgery, GI cancer, immunosuppressive therapy for non-SLE conditions, coexisting autoimmune diseases, pregnancy or lactation, or any current active infection other than H. pylori at enrollment are excluded . Of those eligible, the expected sample size is 115 patients, calculated to power the main outcome analysis. Demographic details (age, sex, ethnicity, disease duration, smoking status, and family history) and clinical manifestations (SLE-related symptoms, medications, and organ involvement) will be thoroughly documented to ensure a well-characterized, representative population .
Sampling Method: Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2026-08-30 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Association between H. pylori infection status and SLE disease activity | baseline
  The study will determine whether the presence or absence of H. pylori infection (measured by stool antigen test) is linked to higher disease activity in SLE, as quantified by the SLEDAI-2K score

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dai X, Fan Y, Zhao X. Systemic lupus erythematosus: updated insights on the pathogenesis, diagnosis, prevention and therapeutics. Signal Transduct Target Ther. 2025 Mar 17;10(1):102. doi: 10.1038/s41392-025-02168-0. PMID 40097390